CLINICAL TRIAL: NCT04978805
Title: The Effect of Progressive Relaxation Exercise on Dyspnea, Pain and Sleep Quality in Lung Cancer Patients Receiving Chemotherapy
Brief Title: Progressive Relaxation Exercise on Dyspnea, Pain and Sleep Quality
Acronym: Progressive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, PhD., Assistant Prof, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/03 - 27
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Cancer
Keywords: Cancer patients; Pain; Sleep quality; Progressive Relaxation Exercise
MeSH Terms: conditions — Neoplasms; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test contro
Who Masked: Participant
Masking Description: Progressive Relaxation Exercise and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Relaxation Exercise (Experimental): A total of 56 sessions of progressive relaxation were performed, 7 days a week for 8 weeks. Each session is set as fifty minutes
  Interventions: Behavioral: Progressive Relaxation Exercise
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercise — In the progressive relaxation technique, the tension and anxiety in skeletal muscles are relatively relieved.
  Arms: Progressive Relaxation Exercise

SUMMARY:
This study was planned to examine the effect of progressive relaxation exercises applied to lung cancer patients receiving chemotherapy on dyspnea, pain and sleep quality.

DETAILED DESCRIPTION:
It is thought that relaxation exercises reduce respiratory distress and improve sleep quality in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65
* Ability to communicate adequately
* Absence of psychiatric problems
* Those who are determined by the physician that they do not have a physical disability in exercising
* Volunteering to participate in the research
* Individuals who have the ability to use technological tools
* Patients with at least 3 cures

Exclusion Criteria:

* Individuals with phones that do not have voice recording capabilities
* Individuals with phones that do not have the ability to install Whatsapp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Visual Analog Scale | 4. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Visual Analog Scale | 8. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Pittsburgh Sleep Quality Index (PSQI) | 1.week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"
Pittsburgh Sleep Quality Index (PSQI) | 4.week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"
Pittsburgh Sleep Quality Index (PSQI) | 8.week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"
Modified Medical Research Council (mMRC) | 1.week
  It is a 5-item scale developed by English Medical Research Council to evaluate dyspnea. While applying Medical Research Council Dyspnea Scale, the patients are asked to indicate the level of activity that creates dyspnea in them. The patient chooses the most appropriate level that defines the respiratory problem by reading the options in the scale. The options are scored between 0 and 4; 0 means no dyspnea, 1 means mild dyspnea (respiratory distress when moving quickly and climbing slightly uphill); 2 means moderate dyspnea (walking slower than peers when walking straight on, stopping to breathe); 3 means severe dyspnea (stopping to breathe after walking about 100 m or for a few minutes) and 4 means very severe dyspnea (getting out of breath while doing daily chores at home, while putting on and taking off clothes and while going to toilet).
Modified Medical Research Council (mMRC) | 4.week
  It is a 5-item scale developed by English Medical Research Council to evaluate dyspnea. While applying Medical Research Council Dyspnea Scale, the patients are asked to indicate the level of activity that creates dyspnea in them. The patient chooses the most appropriate level that defines the respiratory problem by reading the options in the scale. The options are scored between 0 and 4; 0 means no dyspnea, 1 means mild dyspnea (respiratory distress when moving quickly and climbing slightly uphill); 2 means moderate dyspnea (walking slower than peers when walking straight on, stopping to breathe); 3 means severe dyspnea (stopping to breathe after walking about 100 m or for a few minutes) and 4 means very severe dyspnea (getting out of breath while doing daily chores at home, while putting on and taking off clothes and while going to toilet).
Modified Medical Research Council (mMRC) | 8.week
  It is a 5-item scale developed by English Medical Research Council to evaluate dyspnea. While applying Medical Research Council Dyspnea Scale, the patients are asked to indicate the level of activity that creates dyspnea in them. The patient chooses the most appropriate level that defines the respiratory problem by reading the options in the scale. The options are scored between 0 and 4; 0 means no dyspnea, 1 means mild dyspnea (respiratory distress when moving quickly and climbing slightly uphill); 2 means moderate dyspnea (walking slower than peers when walking straight on, stopping to breathe); 3 means severe dyspnea (stopping to breathe after walking about 100 m or for a few minutes) and 4 means very severe dyspnea (getting out of breath while doing daily chores at home, while putting on and taking off clothes and while going to toilet).

CONTACTS AND LOCATIONS:
Locations (1):
- Zülfünaz, Istanbul, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borji M, Nourmohammadi H, Otaghi M, Salimi AH, Tarjoman A. Positive Effects of Cognitive Behavioral Therapy on Depression, Anxiety and Stress of Family Caregivers of Patients with Prostate Cancer: A Randomized Clinical Trial. Asian Pac J Cancer Prev. 2017 Dec 28;18(12):3207-3212. doi: 10.22034/APJCP.2017.18.12.3207. PMID 29281868
- [Background] Tsitsi T, Charalambous A, Papastavrou E, Raftopoulos V. Effectiveness of a relaxation intervention (progressive muscle relaxation and guided imagery techniques) to reduce anxiety and improve mood of parents of hospitalized children with malignancies: A randomized controlled trial in Republic of Cyprus and Greece. Eur J Oncol Nurs. 2017 Feb;26:9-18. doi: 10.1016/j.ejon.2016.10.007. Epub 2016 Nov 18. PMID 28069156
- [Derived] Turan GB, Ozer Z, Sarikose A. The effects of progressive muscle relaxation exercise applied to lung cancer patients receiving chemotherapy on dyspnea, pain and sleep quality: A randomized controlled trial. Eur J Oncol Nurs. 2024 Jun;70:102580. doi: 10.1016/j.ejon.2024.102580. Epub 2024 Apr 1. PMID 38636116